CLINICAL TRIAL: NCT02373605
Title: Spinal Manipulation and Dry Needling Versus Conventional Physical Therapy in Patients With Cervicogenic Headache: a Multi-center Randomized Clinical Trial
Brief Title: Spinal Manipulation and Dry Needling Versus Conventional Physical Therapy in Patients With Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, DPT MSc FAAOMPT, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0001
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Cervicogenic Headaches
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Dry Needling; Manipulation, Spinal; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Needling,Thrust Manipulation (Experimental)
  Interventions: Other: Dry Needling,Thrust Manipulation
- Exercise,Non-thrust Mobilization (Active Comparator)
  Interventions: Other: Exercise,Non-thrust Mobilization

INTERVENTIONS:
Other: Dry Needling,Thrust Manipulation — HVLA thrust manipulation to upper cervical and upper thoracic regions. Dry needling to cervicothoracic and craniofacial regions. Up to 8 treatment sessions over 4 weeks.
  Other Names: Spinal Manipulation; Dry Needling
  Arms: Dry Needling,Thrust Manipulation
Other: Exercise,Non-thrust Mobilization — Non-thrust mobilization and exercise to upper cervical and upper thoracic regions. Up to 8 treatment sessions over 4 weeks.
  Other Names: Exercise; Non-thrust Mobilization
  Arms: Exercise,Non-thrust Mobilization

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with cervicogenic headaches: non-thrust mobilization and exercise versus thrust manipulation and dry needling. Physical therapists commonly use all of these techniques to treat cervicogenic headaches. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with cervicogenic headaches will be randomized to receive 1-2 treatment sessions per week for 4 weeks (up to 8 sessions total) of either: (1) Dry Needling and HVLA thrust manipulation group, or the (2) Exercise and non-thrust mobilization group

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cervicogenic headache as defined by Cervicogenic Headache International Study Group criteria
2. Headache frequency of at least one per week for a minimum of 3 months
3. Minimum pain score (NPRS) of 2/10 and minimum disability score (NDI) of 10/50

Exclusion Criteria:

1. Presence of any of the following atherosclerotic risk factors: hypertension, diabetes, heart disease, stroke, transient ischemic attack, peripheral vascular disease, smoking, hypercholesterolemia or hyperlipidemia
2. Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e. tumors, fracture, metabolic diseases, RA, osteoporosis, history of prolonged steroid use, etc.
3. History of whiplash injury within the last 6 weeks
4. Diagnosis of cervical stenosis
5. Bilateral upper extremity symptoms
6. Evidence of CNS involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes).
7. Two or more positive neurologic signs consistent with nerve root compression, including any 2 of the following:

   1. Muscle weakness involving a major muscle group of the upper extremity.
   2. Diminished UE deep tendon reflex of the biceps, brachioradialis, triceps or superficial flexors
   3. Diminished or absent sensation to pinprick in any UE dermatome.
8. Prior surgery to neck of thoracic spine
9. Involvement in litigation or worker's compensation regarding their neck pain and/or headaches
10. PT or chiropractic care treatment for neck pain or headaches in the 3 months prior to baseline exam.
11. Any condition that might contraindicate spinal manipulative therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-02; Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Headache Intensity (NPRS) (Rating Score) | Baseline, 1 week, 4 weeks, 3 months
  Rating Score. Baseline score must exceed 2/10 to be included in the study.
Change in Headache Frequency (Number of headaches in the last week) | Baseline, 1 week, 4 weeks, 3 months
  Number of headaches in the last week
Change in Disability (NDI 0-50 points) | Baseline, 1 week, 4 weeks, 3 months
  10 Questions each worth 0-5 points with maximum score of 50 points possible. Baseline score must exceed 10/50 to be included in study.

SECONDARY OUTCOMES:
Change in Global Rating of Change Score | 1 week, 4 weeks, 3 months
Change in Medication Intake (Frequency of medication intake in last week) | Baseline, 3 months
Change in Headache Duration (Total hours of headaches in the last week) | Baseline, 1 week, 4 weeks, 3 months
  Total hours of headaches in the last week

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT PhD, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Alabama Physical Therapy & Acupuncture, Montgomery, Alabama, United States

REFERENCES:
- [Derived] Dunning J, Butts R, Zacharko N, Fandry K, Young I, Wheeler K, Day J, Fernandez-de-Las-Penas C. Spinal manipulation and perineural electrical dry needling in patients with cervicogenic headache: a multicenter randomized clinical trial. Spine J. 2021 Feb;21(2):284-295. doi: 10.1016/j.spinee.2020.10.008. Epub 2020 Oct 13. PMID 33065273